CLINICAL TRIAL: NCT06569706
Title: Feasibility and Acceptability of Endoscopic Mastectomy in Patients With Breast Cancer
Acronym: NEOMAMENDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24_0132_UF7830; 2024-A01008-39 (Other: ID-RCB)
Record Dates: First submitted 2024-08-13; First posted 2024-08-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Subcutaneous Mastectomy; Endoscopy; Breast reconstruction; Breast implants; Cancer patients
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nipple-Sparing Mastectomy, with immediate breast reconstruction (Experimental): 20 patients female with breast cancer will have a Nipple-Sparing Mastectomy, with immediate breast reconstruction
  Interventions: Procedure: Nipple-Sparing Mastectomy, with immediate breast reconstruction

INTERVENTIONS:
Procedure: Nipple-Sparing Mastectomy, with immediate breast reconstruction — It is an endoscopic approach for mastectomy using an axillary single port
  Other Names: Endoscopic approach of nipple-sparing mastectomy, with immediate breast reconstruction

SUMMARY:
Nipple -Sparing Mastectomy (NSM), with immediate breast reconstruction (IBR) can be offered to patients requiring mastectomy when the lesion is more than 2cm from the nipple. Endoscopic mastectomy is a technical alternative for small-volume breasts (cup sizes A, B, C), offering a NSM with IBR, but also concealing the scar on the axillary line. It can be performed with traditional laparoscopic equipment, making this technique much more accessible and less costly than robotic mastectomy. It uses a single-port device that is significantly less costly than robotic equipment.

Feasibility and safety studies remain limited to the Asian continent, and it would undoubtedly be beneficial to initiate research in Europe to add this new technical option to our surgical arsenal. This study project aims to explore the feasibility and safety of endoscopic nipple-sparing mastectomy for breast cancer indications in a French center.

DETAILED DESCRIPTION:
It s a practicability study, evaluating endoscopic approach for mastectomy, using an axillary single port in breast cancer patients. Conventional surgery conversion rate, operative time, infectious rate, esthetical outcomes, oncological safety and functional outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20 and 75 years.
* Patient with an indication for curative mastectomy, either unilateral or bilateral, with nipple preservation:

  * Extensive Carcinoma In Situ (CIS), more than 2 cm from the nipple
  * Multicentric Infiltrating Carcinoma (IC), more than 2 cm from the nipple
  * Large volume Infiltrating Carcinoma, more than 2 cm from the nipple
  * IC or CIS for which the patient refuses conservative treatment, more than 2 cm from the nipple
* Breast volumes: cup sizes A, B, or C as defined by underwear size, and glandular ptosis not exceeding grade 2 according to Regnault's classification
* Patient wishing to undergo immediate breast reconstruction.
* WHO/OMS (World Health Organization/Organisation Mondiale de la Santé) performance status <3

Exclusion Criteria:

* Cutaneous carcinoma
* Inflammatory breast
* History of oncological breast surgery on the same breast
* Patient who has received radiation treatment on the same breast
* Breast hypertrophy requiring a nipple-bearing flap
* Smoking ≥ 10 cigarettes/day
* BMI > 35
* Protected patient or unable to give consent according to Article L1121-8 of the French Public Health Code (CSP).
* Patient participating in another interventional clinical study.
* ASA (physical status score of the American Society of Anesthesiologists) >2.
* Pregnant or breastfeeding women according to Article L1121-5 of the CSP.
* Vulnerable persons (those receiving psychiatric care, those deprived of liberty, and those admitted to a health or social institution) according to Article L1121-6 of the CSP.
* Absence of effective contraception for patients of childbearing age.
* Absence of affiliation with a social security scheme.
* Absence of collected free, informed, and written consent.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2029-10-18 (Estimated)

PRIMARY OUTCOMES:
Success rate of endoscopic nipple sparing mastectomy (E-NSM) for breast cancer patients. | one day
  The E-NSM is done by a scar in the axillary area, away from the breast, using single port endoscopy, with Implant base reconstruction in pre pectoral position.
  - Complete excision of the gland by means of an incision on the axillary line, installation of a definitive smooth prosthesis, absence of conversion to a conventional approach.

SECONDARY OUTCOMES:
Operative time | one day
  Duration of the prophylactic mastectomy with immediate breast reconstruction
Hospital stay | Through discharge from hospitalization, an average of 7 days
  The duration of hospitalization will be noted upon discharge from hospitalization
Open surgery conversion rate | one day
  Number of patients with open surgery conversion
Oncologic safety of this approach | 1 and 2 years after surgery
  Evaluation of the early local recurrence of breast cancer rate at 1 and 2 year by imaging (breast ultrasound and/or MRI) and clinical examination.
  Recurrence will be defined by an attenuating tissue mass on ultrasound and/or suspicious contrast on MRI and/or a clinically palpable nodule, that will be confirmed by biopsy with histological analysis.
Concealed nature of the breast scar | Before surgery and 1 month and 3 months after surgery
  Number of patients with no visible scars, picture taken bare chest front and side after the surgery
Number of participants with an infection | At surgery, and 1, 3, months after surgery
  Number of participants with postoperative infection after the mastectomy, including cases requiring implant replacement or removal.
Skin case necrosis | At surgery, and 1, 3, 6, 12, 18, and 24 months after surgery
  The presence of skin case necrosis will be noted during all the visits after the surgery. It's severe if > 25%
Complication rates (ischemia) | At surgery, and 1, 3, 6, 12, 18, and 24 months after surgery
  Nipple-Areola-Complex (NAC) Ischemia: comparison with literature data on conventional surgery, including grading of ischemia
Number of participants with a local haematoma | At surgery, and 1, 3, 6, 12, 18, and 24 months after surgery
  Number of participants with a local haematoma caused by the mastectomy with immediate breast reconstruction requiring surgical intervention.
Post-operative seromas | At surgery, and 1, 3, 6, 12, 18, and 24 months after surgery
  Number of patients with seromas after the mastectomy
Necrosis of areolo-nipple plaque | At surgery, and 1, 3, 6, 12, 18, and 24 months after surgery
  The presence of necrosis of areolo-nipple plaque will be noted during all the visits after the surgery.
Aesthetic result | 90 days and 1 year after surgery
  BREAST-Q© questionnaire Version 1.0 measure the quality of life and satisfaction among patients undergoing breast surgery. This questionnaire includes 6 modules: 1) Augmentation module, 2) Reduction/Mastectomy module, 3) Breast cancer: a) Mastectomy module, b) Reconstruction module, c) Breast reconstruction expectations module, d) Breast conserving therapy module.
  The conceptual framework of the modules is comprised of following two overarching themes (or domains): 1) Health-related quality of life and 2) Patient satisfaction. 1) Under each of these domains, there are six subthemes; Quality of life: 1) Psychosocial, 2) Physical and 3) Sexual well-being; and Patient satisfaction: 4) Satisfaction with Breasts, 5) Satisfaction with Outcome and 6) Satisfaction with care.
  Cf. https://qportfolio.org/wp-content/uploads/2023/01/BREAST-Q-BREAST-CANCER-USER-GUIDE.pdf for the response options.
Life quality | Before surgery and 90 days and 1 year after surgery
  Quality of life with an european quality of life scale (EQ-5D-5L). The EQ-5D-5L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, few problems, some problems, severe problems and extreme problems. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having few problems for 2, some problems for 3, severe problems for 4, and having extreme problems for 5. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 55555 (having extreme problems in all dimensions).

CONTACTS AND LOCATIONS:
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No